CLINICAL TRIAL: NCT03939949
Title: Mindfully Attending to Pain Sensations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Karyn Gunnet-Shoval, Co-Investigator, Harvard University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB17-1861
Record Dates: First submitted 2019-02-09; First posted 2019-05-07 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
Keywords: pain; mindfulness; awareness; attention to variability; quality of life; wellbeing
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware of how the conditions differ, nor are they aware of how many conditions there are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Mindfulness (Experimental): All participants in this condition will complete all measures online at four different points in time, including one narrative response at T1. They will also be instructed to complete a mindfulness intervention at home and respond to diary-type text messaging questions (all including questions about pain) twice daily for six days.
  Interventions: Behavioral: High Mindfulness
- Low Mindfulness (Experimental): All participants in this condition will complete all measures online at four different points in time, including one narrative response at T1. They will also be instructed to respond to diary-type text messaging questions (some related to pain) twice daily for six days.
  Interventions: Behavioral: Low Mindfulness
- Active control (Active Comparator): All participants in this condition will complete all measures online at four different points in time, including one narrative response at T1. They will also be instructed to respond to diary-type text messaging questions (none about pain) twice daily for six days.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: High Mindfulness — Those in the "high mindfulness" group will also receive questions about their current pain intensity and unpleasantness in both the morning and evening for six days. In order to emphasize the variability in pain, participants will receive these text messages on a variable schedule. In addition, they will sent instructions every morning to pay attention to variability in their pain throughout the day and asked to report on how their pain is changing over time as a part of each text message prompt.
  Arms: High Mindfulness
Behavioral: Low Mindfulness — Those in the "low mindfulness" group, who will receive receive two text messages per day (one at at 9am and one at 9pm) for six days, each prompting them to write about the activity they are currently engaged in. They will also be prompted with the 9pm text to report on their pain intensity and unpleasantness at that time.
  Arms: Low Mindfulness
Behavioral: Active Control — Participants in the "active control" group will receive 2 text messages per day for six days (one at 9am and one at 9pm) asking them to report on the activity they are currently engaged in.
  Arms: Active control

SUMMARY:
Substantial evidence suggests that psychosocial factors play a key role in explaining the risk for development of chronic pain, as well as for coping with it. Such factors include psychological perceptions or orientation towards pain, mainly referring to fear of pain and pain catastrophizing. Nonetheless, although this link is well documented, the underlying mechanisms of these processes have yet to be established. The "Attention to Variability" paradigm presents an explanatory mechanism, according to which the ability to mindfully attend to chronic symptoms enables and promotes increased control over the etiology and the expression of chronic symptoms. In support of the ATV paradigm, empirical findings demonstrate that ATV improved pregnancy outcomes and allowed people to gain control over fluctuations in their heart rates.

The goal of the present study is to examine whether mindfully attending to pain sensations will decrease the intensity and frequency of chronic pain, increase perceived control of pain, and improve well-being and health-related quality of life.

DETAILED DESCRIPTION:
Participants who experience chronic pain will be randomly assigned to one of three experimental groups, which differ in the content and scheduling of text messages delivered over a period of six days. One third of participants will be assigned to the "active control" group. These participants will receive 2 text messages per day for six days (one at 9am and one at 9pm) asking them to report on the activity they are currently engaged in. One third of participants will be assigned to the "low mindfulness" group. These participants will receive the same text messages as the participants in the active control group, but will also be prompted with the 9pm text to report on pain intensity and unpleasantness at that time. One third of participants will be assigned to the "high mindfulness" group. These participants will also receive two text message prompts about their current activity. Participants in the "high mindfulness" group will also receive questions about current pain intensity and unpleasantness in both the morning and evening. In order to emphasize the variability in pain, participants will receive these text messages on a variable schedule. In addition, they will sent instructions every morning to pay attention to variability in their pain throughout the day and asked to report on how their pain is changing over time as a part of each text message prompt.

The researchers will take measurements of pain interference, perceptions of control, and pain experience at three time points (T0=baseline, T1= immediately after the 6 days of text messages, T2= 1 month after T1, and T3= 3 months after T1). All surveys will be collected online via the Qualtrics.com platform.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Suffer from chronic pain (at least six months)
* Evaluate their usual level of pain in the last week as 4 and above (on a numeric rating scale from 0-10 with 0 indicating "No Pain" and 10 indicating "Worst pain imaginable)
* Fluent in English
* Owns a smartphone

Exclusion Criteria:

* Individuals under the age of 18;
* Individuals who are not patients of our collaborating pain clinics or online chronic pain support groups and/or do not endorse their pain as chronic.
* Individuals who are pregnant
* Individuals with diagnosed cognitive impairment
* Individuals who would not be able to read text messages because of visual impairment
* Individuals with ongoing/current complications from spinal cord injury
* Individuals with active cancer
* Amputees
* Individuals with unhealed fractures
* Diabetics who do not have symptoms under control
* Individuals who have visited a doctor for a fall in the last 6 months
* Individuals with the diagnosis of schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Beliefs and Perceptions Inventory (PBAPI) | 2 minutes
  The objective of the measure is to assess new pain believes. The scale includes 16 questions, each ranging from -2 to 2, with -2 being 'Strongly Disagree' and 2 being 'Strongly Agree.' There is no zero point on the scale. The 16-question measure includes four subscales, each containing four items. The subscales (Pain as Mystery, Pain as Constant, Pain as Permanent and Self-Blame) are scored individually by adding the score for each of the four items within a subscale together and then dividing that number by four. The subtotal for each one is then added to the others for a total scale score. Five items are reverse-scores, two of which are in the Pain as Constant subscale and the other three of which are in the Pain as Permanent Subscale. Final scores can range from -8 to 8.
Multidimensional Health Locus of Control Scale - Form C (MHLC-Form C) | 3 minutes
  The objective of the assessment is to measure health-related control beliefs in individuals with an current medical condition, such that scoring indicate the degree to which an individual believes their health is under their control versus the control of others or external forces. The scale includes 18 items, each ranging from 1-6, with 1 being 'Strongly Disagree' and 6 being 'Strongly Agree'. The scale includes four subscales including Internal, Chance, Doctors, and Other People. To determine overall scale score, sum all items from all subscales together for a final score between 18 and 108.
Brief Pain Inventory- Short Form | 2 minutes
  9-item scale measures pain severity and impact of pain on functional health. First item asks whether they have pain other than 'everyday' pain today (yes/No). Second question provides diagram of a person, asking one to point to pain and most pain. Next four items ask one to rate the worst, least, average and current pain over past 24 hours on a scale from 0 (No Pain)-10 (Pain As Bad As You Can Imagine). Item 7 asks about current pain treatments. Item 8 asks about % relief pain treatments provided over last 24 hours. %'s range from 0 (No Relief) to 100 (Complete Relief). Last item asks one to indicate pain interfering with 'General Activity,' 'Mood,' 'Walking ability,' 'Normal work,' 'Relations with other people,' 'Sleep,' and 'Enjoyment of life' over past 24 hours. Scales range from 0 (Does Not Interfere) to 10 (Completely Interferes). A mean composite score of items 3-6 yields pain severity. Other items are to be individually interpreted.
The MOS 36-Item Short-Form Health Survey (SF-36) | 3 minutes
  The objective of the measure is to survey health status. The assessment includes 36 items, with eight scaled scores from 8 separate dimensions, including 'Vitality,' 'Physical Functioning,' 'Bodily Pain,' 'General Health Perceptions,' 'Physical Role Functioning,' 'Emotional Role Functioning,' 'Social Role Functioning' and 'Mental Health.' Scores range from 0-100 with lower scores indicating more disability and higher score indicating less disability.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | 2 minutes
  The objective of the assessment is to measure catastrophic thinking related to pain. The tool asks individuals to endorse the degree to which they identified with certain thoughts or emotions surrounding their previous experiences of pain. The measure includes 13 items asking participants to rate their responses on a five-point likert scale ranging from 0 (not at all) to 4 (all the time). The measure consists of three subscales, including 'Rumination', 'Magnification' and 'Helplessness.' To score the measure, one is to sum up each of the subscales and then calculate the sum of the three subscales together. The subscales can also be individually interpreted.
Langer Mindfulness Scale- 14 item (LMS-14) | 2 minutes
  The assessment measures socio-cognitive mindfulness. The measure includes three subscales, each ranging from 1-7, with 1 being 'Strongly Disagree' and 7 being 'Strongly Agree'. Subscales are 'Novelty Seeking'; 'Novelty Producing'; 'Engagement'. Some items are reverse scored. To determine overall Mindfulness score, sum all items (items 1-14).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bercovitz, MA, Principal Investigator — Harvard University; Karyn Gunnet-Shoval, PhD, Principal Investigator — Harvard University; Ellen Langer, PhD, Study Director — Harvard University
Locations (4):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard University, Cambridge, Massachusetts
  - New England Physiatry, Stoneham, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crombez G, Vlaeyen JW, Heuts PH, Lysens R. Pain-related fear is more disabling than pain itself: evidence on the role of pain-related fear in chronic back pain disability. Pain. 1999 Mar;80(1-2):329-39. doi: 10.1016/s0304-3959(98)00229-2. PMID 10204746
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Langer E, Drinka PJ, Voeks SK. Estimating nutritional intake in nursing home residents. Wis Med J. 1989 Dec;88(12):23-5. No abstract available. PMID 2618067
- [Background] Zilcha-Mano S, Langer E. Mindful Attention to Variability Intervention and Successful Pregnancy Outcomes. J Clin Psychol. 2016 Sep;72(9):897-907. doi: 10.1002/jclp.22294. Epub 2016 Mar 23. PMID 27007939
- [Background] Edwards RR, Dworkin RH, Sullivan MD, Turk DC, Wasan AD. The Role of Psychosocial Processes in the Development and Maintenance of Chronic Pain. J Pain. 2016 Sep;17(9 Suppl):T70-92. doi: 10.1016/j.jpain.2016.01.001. PMID 27586832
- [Background] Tsur N, Defrin R, Ginzburg K. Posttraumatic Stress Disorder, Orientation to Pain, and Pain Perception in Ex-Prisoners of War Who Underwent Torture. Psychosom Med. 2017 Jul/Aug;79(6):655-663. doi: 10.1097/PSY.0000000000000461. PMID 28658194
- See also: Additional Reference — https://www.researchgate.net/publication/38413929_The_Effect_of_Mindfulness_on_Heart_Rate_Control

DOCUMENTS (1):
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03939949/ICF_000.pdf